CLINICAL TRIAL: NCT00378768
Title: A Phase II Study of Thymoglobulin in Patients With Multiple Myeloma Who Are Candidates for Allogeneic or Autologous Stem Cell Transplant
Brief Title: Antithymocyte Globulin in Treating Patients Undergoing Stem Cell Transplant for Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 2029.00; FHCRC-2029.00; GENZ-FHCRC-2029.00; CDR0000500474 (Registry Identifier: PDQ)
Record Dates: First submitted 2006-09-19; First posted 2006-09-21 (Estimated); Last update posted 2011-11-30 (Estimated); Status verified 2011-11

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Antilymphocyte Serum

INTERVENTIONS:
Biological: anti-thymocyte globulin

SUMMARY:
RATIONALE: Biological therapies, such as antithymocyte globulin, may stimulate the immune system in different ways and stop cancer cells from growing.

PURPOSE: This phase II trial is studying how well antithymocyte globulin works in treating patients undergoing stem cell transplant for multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate at 4 weeks in patients with multiple myeloma treated with anti-thymocyte globulin at least 4 to 6 weeks prior to undergoing conditioning therapy for allogeneic or autologous stem cell transplantation.

Secondary

* Determine the toxicity of this drug, in terms of formation of antirabbit antibodies, in these patients.

OUTLINE: This is an open-label, multicenter study.

Patients receive anti-thymocyte globulin IV over 6 hours on day 1 and over 4 hours on days 3 and 5. Treatment begins 4 to 6 weeks prior to undergoing conditioning therapy for autologous or allogeneic stem cell transplantation.

After completion of study treatment, patients are followed at 28 days.

PROJECTED ACCRUAL: A total of 12 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed multiple myeloma
* Candidate for autologous or allogeneic stem cell transplantation within 1 to 3 months after study treatment
* Measurable disease, defined as serum monoclonal protein ≥ 1 g/dL OR urinary light chain excretion = 500 mg/24 hours
* No malignant CNS disease

PATIENT CHARACTERISTICS:

* Life expectancy ≥ 6 months
* Absolute neutrophil count ≥ 1,000/mm³
* Platelet count > 50,000/mm³
* Creatinine ≤ 2 mg/dL
* Hepatic function ≤ 2 times upper limit of normal
* DLCO ≥ 50%
* No active infection
* No hypersensitivity to rabbit proteins
* No symptomatic hyperviscosity syndrome
* Negative pregnancy test

PRIOR CONCURRENT THERAPY:

* More than 28 days since prior chemotherapy, including prednisone (20 mg equivalent/day)
* No prior anti-thymocyte globulin
* No concurrent radiotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2005-11; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Response rate, as measured by International Bone Marrow Transplant Registry (IBMTR)/European Group for Blood and Marrow Transplantation (EBMT) Response Criteria, at 4 weeks

SECONDARY OUTCOMES:
Toxicity as assessed by NCI CTC v2.0
Formation of antirabbit antibodies

CONTACTS AND LOCATIONS:
Overall Officials: William I. Bensinger, MD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States